CLINICAL TRIAL: NCT06611865
Title: Cross-sectional Study Documenting the Relative Efficacy of Intraligamentary Anesthesia and the Inferior Alveolar Nerve Block for the Extraction of Posterior Mandibular Teeth.
Brief Title: Comparison of Intraligamentary Anesthesia With the Inferior Alveolar Nerve Block for the Extraction of Mandibular Molars.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamza Zia Ahmed (Other)
Responsible Party: Sponsor-Investigator, Hamza Zia Ahmed, Principal Investigator, Nishtar Medical University
Organization: Nishtar Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 642/NID
Record Dates: First submitted 2024-09-15; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Tooth Extraction; Tooth Extraction Site Healing
Keywords: Intraligamentary Anaesthesia; Inferior Alveolar Nerve Block; Tooth Extraction; Dry Socket
MeSH Terms: conditions — Dry Socket

STUDY DESIGN:
Intervention Model Description: A split-mouth group was included with 70 teeth extracted from 35 patients. In such cases, involving bilaterally indicated teeth, ILA and IANB were used on opposite sides, but the second tooth was anesthetized only after the first extraction had completed and had been recorded. The second group had 500 patients with unilateral extractions. ILA was compared with IANB in each group separately, and the results in group I were then compared descriptively with those in group II.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Split-mouth group (Active Comparator): It includes bilaterally indicated teeth. ILA and IANB were used on opposite sides in the same person; the second tooth was anesthetized only after the first extraction had completed and had been recorded.
  Interventions: Procedure: Intraligamentary anaesthesia; Procedure: Inferior alveolar nerve block
- Group 2 ILA (Active Comparator): The patients in group 2, with unilateral extractions, that were only administered Intraligamentary anaesthesia.
  Interventions: Procedure: Intraligamentary anaesthesia
- Group 2 IANB (Active Comparator): The patients in group 2, with unilateral extractions, that were only administered the Inferior Alveolar Nerve Block. In case of multiple unilaterally indicated teeth that were to be extracted under IANB, only the tooth best fitting all criteria was considered for the study.
  Interventions: Procedure: Inferior alveolar nerve block

INTERVENTIONS:
Procedure: Intraligamentary anaesthesia — Injection of anesthetic solution into the intraligamentary space along the long axis of a tooth root using a pressure syringe.
  Arms: Group 2 ILA; Split-mouth group
Procedure: Inferior alveolar nerve block — Anaesthetic injection into the pterygomandibular space to block the Inferior alveolar nerve at the mandibular foramen point.
  Arms: Group 2 IANB; Split-mouth group

SUMMARY:
Local anaesthesia or numbing is done before tooth extraction. This study compares two different methods of numbing molar teeth before extraction. It compares them on the basis of pain during the procedure and on discomfort after the procedure as well. It will help dentists better understand the benefits of the two techniques, and their usage case to case.

DETAILED DESCRIPTION:
The study was designed as a randomized controlled trial. The purpose of this study was to examine the differences in efficacy of the intraligamentary anaesthetic technique and the inferior alveolar nerve block for mandibular posterior tooth extraction cases. Pain intensity, duration of anaesthesia, incidence of post-operative dry socket, success rates, onset of anaesthesia were examined. It was done in a split-mouth method so that two different techniques were used in the same patient, thus minimizing individual variations.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes who were more than 18 years of age; they had indications of non-surgical extraction of one or multiple mandibular posterior teeth.

Exclusion Criteria:

* For patients: pregnancy, immunological compromise, systemic conditions requiring special considerations and non-compliance.
* The exclusion criteria for individual teeth were: acutely infected teeth or any teeth with the instances of expression of pus through sinus tracts or the gingival sulcus were excluded. In case of multiple unilaterally indicated teeth that were to be extracted under IANB, only the tooth best fitting all criteria was considered for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Injection pain | Through the duration of injection (within a few seconds to 1 minute)
  Rating of injection administration pain from 0-10.
Pain during extraction procedure | For the duration of treatment (estimated within 1 hour)
  Pain during extraction procedure on a scale of 0-10.
Unpleasantness of treatment | For the duration of treatment (estimated within 1 hour)
  A rating of 0-10 for overall discomfort felt by the patient during the treatment.
Latency time of anesthesia (minutes) | Anesthesia was tested with a dental probe on the marginal gingiva at: 1) immediately after the injection and 2) every 10 seconds (ILA) / every 30 seconds (IANB) until complete painlessness was achieved.
  The onset of anesthesia after injection
Anesthetic effect | For the duration of treatment (estimated within 2 hours)
  4 categories: Complete, sufficient, insufficient or no effect.
Amount of anesthetic solution (mL) | For the duration of treatment (estimated within 1 hour)
  The average amount of anaesthetic solution injected per procedure.
Duration of treatment (minutes) | For the duration of treatment (estimated up to 1 to 2 hours)
  Time in minutes taken from the injection to the complete extraction of tooth.
Duration of local numbness (minutes) | For the duration of treatment (estimated up to 1 to 2 hours)
  Total duration of local numbness reported by the patient

SECONDARY OUTCOMES:
Incidence of Dry socket | From the complete extraction of tooth to 14 days after the extraction of tooth
  Dry socket incidence reported by the patient int he recovery period of 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Amjad Bari, MDS, Study Chair — Nishtar Medical University
Locations (1):
- Nishtar Institute of Dentistry, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided